CLINICAL TRIAL: NCT03654469
Title: Bronchial Obstruction in Dairy Farmers
Acronym: BPCO Airbag
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC11_8953; 2011-A01010-41 (Other: Id-RCB)
Record Dates: First submitted 2016-09-13; First posted 2018-08-31 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Plasma of patients are collected
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaires and electronic mini-spirometry — prospective screening study based on questionnaires and electronic mini-spirometry (Néo-6(®)) that includes a representative sample of dairy farmers from the departments of Morbihan and Île-et-Vilaine in Brittany

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major public health problem and is expected to become the 3rd leading cause of death globally by 2020.

The main risk factor is tobacco. Tobacco poisoning is found in 80 to 90% of patients with COPD. However, non-smoking COPD is also described, with increasing prevalence figures, particularly related to occupational exposure, especially among farmers.

DETAILED DESCRIPTION:
A prospective screening study based on questionnaires and electronic mini-spirometry (Néo-6®) that includes a representative sample of dairy farmers from the departments of Morbihan and Île-et-Vilaine in Brittany.

The dairy farmers had an occupational medicine appointment and, if they demonstrated at least one marker of possible bronchial obstruction (chronic cough, chronic bronchitis, dyspnoea, wheezing, spirometry), they were referred to a pulmonologist.

ELIGIBILITY:
Inclusion Criteria:

* dairy farmers from the departments of Morbihan and Île-et-Vilaine in Brittany
* control: non farmer

Exclusion Criteria:

* pigs or grain farmers
* Pregnant women
* oral corticosteroids or immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * dairy farmers from the departments of Morbihan and Île-et-Vilaine in Brittany
  * control: non farmer
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Level of bronchial obstruction | 3 years
  Respiratory specific indices are extracted from a screening spirometry :
  Forced expiratory volume in one second (FEV1) Forced Vital Capacity (FVC)
  Bronchial obstruction is stated with a ratio FEV1 / FVC < 0.8

SECONDARY OUTCOMES:
Prevalence of occupational specific COPD in dairy farmers | 3 years
  Occupational specific COPD is defined as a ratio FEV1 / FVC < 0.8 associated to a clinical situation :
  * non reversibility after β2-agonists or corticoids administration,
  * no personal nor familial allergic conditions,
  * smoking history < 1 cigarettes package per year.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Jouneau, MD, PhD, Study Director — Rennes University Hospital
Locations (1):
- Rennes University Hospital - Service de Pneumologie, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jouneau S, Chapron A, Ropars C, Marette S, Robert AM, Gouyet T, Belleguic C, Rochefort-Morel C, Guillot S, Mailloux C, Desrues B, Viel JF; AIRBAg research group. Prevalence and risk factors of asthma in dairy farmers: Ancillary analysis of AIRBAg. Environ Res. 2022 Nov;214(Pt 4):114145. doi: 10.1016/j.envres.2022.114145. Epub 2022 Aug 20. PMID 35998695